CLINICAL TRIAL: NCT05146947
Title: Intraoperative Near Infrared Spectroscopy of Kidney for Prediction of Acute and Sub-acute Kidney Injury in Partial Nephrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TASMC-21-OG-0327-21-CTIL
Record Dates: First submitted 2021-11-20; First posted 2021-12-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-12

CONDITIONS: Kidney Injury
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: near infrared spectroscopy — near infrared spectroscopy monitoring on kidney after reperfusion

SUMMARY:
Intra-operative NIRS measurements of kidney during partial nephrectomy, after reperfusion, for monitoring ischemia and prediction of postoperative renal dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for partial nephrectomy at Tel Aviv Medical Center who will consent to participate.

Exclusion Criteria:

* Patients unable to give consent,
* Patients who were lost to follow up during the first 7 post-operative days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Acute Kidney Injury | 7 days post operative and during 6 months post-surgery.
  An increase in serum creatinine by 0.3mg/dL or more within 48 hours compared with admission creatinine level or an increase in serum creatinine above 1.5 times baseline within 7 days of admission

SECONDARY OUTCOMES:
Surgical complications | 7 days post operative
  Vascular/Bleeding ect.

CONTACTS AND LOCATIONS:
Overall Officials: Orr Goren, Dr, Principal Investigator — Tel Aviv Medical Center

IPD SHARING:
Plan to Share IPD: No